CLINICAL TRIAL: NCT03157284
Title: Efficacy of Fermented Rice Flour for the Treatment of Atopic Dermatitis : Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Efficacy of Fermented Rice Flour for the Treatment of Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinz Italia SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: FERCT16
Record Dates: First submitted 2017-05-01; First posted 2017-05-17 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Atopic Dermatitis
Keywords: Lactobacillus, Probiotics
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Flour

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo Group will receive 7gr Maltodextrin
  Interventions: Dietary Supplement: Placebo
- Intervention Rice Flour (Experimental): The Intervention Group will receive 7gr of the experimental ingredient fermented Rice Flour
  Interventions: Dietary Supplement: Rice Flour

INTERVENTIONS:
Dietary Supplement: Rice Flour — For 12 weeks, a group of children will receive 7gr fermented rice flour according to a randomised, double-blind design.
  Arms: Intervention Rice Flour
Dietary Supplement: Placebo — For 12 weeks a group of children will receive a 7gr of a placebo (maltodextrin), according to a randomised, double-blind design.
  Arms: Placebo

SUMMARY:
This Study Evaluate the efficacy of the subministration of fermented rice flour (7 g/day) on the clinical course of patients with moderate or severe Atopic Dermatitis, in terms of a reduction in the SCORAD score, during the study period and four weeks after the suspension of the treatment.

DETAILED DESCRIPTION:
It is scientifically recognised that some probiotic effects can be obtained from inactivated bacteria or isolated bacterial components (e.g. bacterial DNA) or factors produced during fermentation (short-chain fatty acids, bacterial proteins, etc.) (7). This category also includes the ingredient which forms the focus of this trial: fermented rice flour, prepared from rice flour fermented by a probiotic (Lactobacillus paracasei CBA L74) which was heat-inactivated at the end of the fermentation process. The finished product, therefore, does not contain live bacteria.

The bacterium used - owned by the sponsor and filed with the BCCM/LMG bacteria collection - belongs to the species Lactobacillus paracasei, and is included in the Qualified Presumption of Safety (QPS) list of microorganisms compiled by the European Food Safety Authority's Panel on Biological Hazards (8). The bacterium has been tested for its sensitivity to antibiotics on the basis of the relevant criteria drawn up by the EFSA (9) and its genomic sequence is known. Pre-clinical studies have shown anti-inflammatory effects of food matrices fermented with Lactobacillus paracasei CBA L74 (stimulating the production of IL-10 and the reduction of IL-12), and in response to stimulation with Salmonella typhimurium (10). Recently, the clinical effects of the consumption of rice flour fermented with Lactobacillus paracasei CBA L74 for 12 weeks were tested in a pilot study conducted on children with moderate/severe AD (defined using the SCORAD index) (11). In this study, all the children reported an improvement in the severity of the AD and reduced topical steroid application frequency.

Considering the rationale for the use of live or inactivated probiotics or isolated bacterial components for the treatment of AD as well as the clinical studies in the paediatric population that have shown encouraging results (11), this randomised, double-blind, placebo-controlled trial aims to evaluate the efficacy of rice flour fermented with Lactobacillus paracasei CBA L74 in subjects with AD; in particular, this trial will evaluate the clinical response in terms of the severity of the AD during and at the end of a 12-week treatment period and four weeks after the suspension of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children between 6 and 36 months old, gradually enrolled from among patients attending the Paediatric Dermatology and Allergy Clinic
* Diagnosis of moderate or severe Atopic Dermatitis, evaluated using the SCORAD index

Exclusion Criteria:

* Rhinitis and/or acute asthma
* Chronic diseases (autoimmune diseases, Cronic Obstructive Pulmunary Disease, heart disease, Congenital Nephrotic diseases, diabetes, acquired or congenital immunodeficiency)
* Treatment with prebiotics and/or probiotics in the month prior to enrolment
* Ongoing antibiotic therapy
* Treatment with systemic immunomodulators in the month prior to enrolment
* Treatment with topical immunomodulators (tacrolimus or pimecrolimus) in the three months prior to enrolment

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-29 (Actual)

PRIMARY OUTCOMES:
Reduction in the SCORAD score | 16 weeks
  Standardised questionnaire for calculating the SCORAD score:
  Evaluate the efficacy of the administration of fermented rice flour (7 g/day) on the clinical course of patients with moderate or severe Atopic Dermatitis, in terms of a reduction in the SCORAD score, during the study period and four weeks after the suspension of the treatment

SECONDARY OUTCOMES:
Inflammatory response :Peripheral immunophenotype analysis and Cytokine profile | 12 weeks
  Evaluate the inflammatory response at baseline (T0) and at the end of treatment (T12) in terms of inflammation markers (cytokine profile) and peripheral immunophenotype compared to the placebo group.Peripheral cytokine assay (IFNγ, IL-4, IL-5, IL-10, IL-12, IL-13, IL-18, IL-31) at baseline and after specific stimulation (anti-CD3/CD28) or non-specific stimulation (PHA) on all enrolled children.
Allergic sensitisation:Total and specific IgE (sIgE) assay | 12 weeks
  Evaluate allergic sensitisation by total and specific IgE (sIgE) assay at baseline (T0) and at the end of treatment (T12) compared to the placebo group
Steroids prescription | 16 weeks
  Evaluate the prescription of topical steroid therapy in the group of children treated with fermented rice flour compared to the placebo group.
Faecal microbiota analysis | 12 weeks
  Evaluate the change in intestinal microbial flora between T0 and T12

CONTACTS AND LOCATIONS:
Overall Officials: EnzaCarmina D'Auria, Dott, Principal Investigator — Clinica Pediatrica Ospedale dei Bambini Vittore Buzzi
Locations (1):
- Ospedale dei Bambini Vittore Buzzi-Clinica Pediatrica, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elias PM, Steinhoff M. "Outside-to-inside" (and now back to "outside") pathogenic mechanisms in atopic dermatitis. J Invest Dermatol. 2008 May;128(5):1067-70. doi: 10.1038/jid.2008.88. PMID 18408746
- [Background] Sidbury R, Tom WL, Bergman JN, Cooper KD, Silverman RA, Berger TG, Chamlin SL, Cohen DE, Cordoro KM, Davis DM, Feldman SR, Hanifin JM, Krol A, Margolis DJ, Paller AS, Schwarzenberger K, Simpson EL, Williams HC, Elmets CA, Block J, Harrod CG, Smith Begolka W, Eichenfield LF. Guidelines of care for the management of atopic dermatitis: Section 4. Prevention of disease flares and use of adjunctive therapies and approaches. J Am Acad Dermatol. 2014 Dec;71(6):1218-33. doi: 10.1016/j.jaad.2014.08.038. Epub 2014 Sep 26. PMID 25264237
- [Background] Isolauri E, Arvola T, Sutas Y, Moilanen E, Salminen S. Probiotics in the management of atopic eczema. Clin Exp Allergy. 2000 Nov;30(11):1604-10. doi: 10.1046/j.1365-2222.2000.00943.x. PMID 11069570
- [Background] Weston S, Halbert A, Richmond P, Prescott SL. Effects of probiotics on atopic dermatitis: a randomised controlled trial. Arch Dis Child. 2005 Sep;90(9):892-7. doi: 10.1136/adc.2004.060673. Epub 2005 Apr 29. PMID 15863468
- [Background] Majamaa H, Isolauri E. Probiotics: a novel approach in the management of food allergy. J Allergy Clin Immunol. 1997 Feb;99(2):179-85. doi: 10.1016/s0091-6749(97)70093-9. PMID 9042042
- [Background] Sistek D, Kelly R, Wickens K, Stanley T, Fitzharris P, Crane J. Is the effect of probiotics on atopic dermatitis confined to food sensitized children? Clin Exp Allergy. 2006 May;36(5):629-33. doi: 10.1111/j.1365-2222.2006.02485.x. PMID 16650048
- [Background] Agostoni C, Goulet O, Kolacek S, Koletzko B, Moreno L, Puntis J, Rigo J, Shamir R, Szajewska H, Turck D; ESPGHAN Committee on Nutrition. Fermented infant formulae without live bacteria. J Pediatr Gastroenterol Nutr. 2007 Mar;44(3):392-7. doi: 10.1097/01.mpg.0000258887.93866.69. PMID 17325568
- [Background] Zagato E, Mileti E, Massimiliano L, Fasano F, Budelli A, Penna G, Rescigno M. Lactobacillus paracasei CBA L74 metabolic products and fermented milk for infant formula have anti-inflammatory activity on dendritic cells in vitro and protective effects against colitis and an enteric pathogen in vivo. PLoS One. 2014 Feb 10;9(2):e87615. doi: 10.1371/journal.pone.0087615. eCollection 2014. PMID 24520333
- [Background] Beretta S, Fabiano V, Petruzzi M, Budelli A, Zuccotti GV. Fermented rice flour in pediatric atopic dermatitis. Dermatitis. 2015 Mar-Apr;26(2):104-6. doi: 10.1097/DER.0000000000000103. No abstract available. PMID 25757084
- [Background] Severity scoring of atopic dermatitis: the SCORAD index. Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology. 1993;186(1):23-31. doi: 10.1159/000247298. PMID 8435513
- [Background] Schram ME, Spuls PI, Leeflang MM, Lindeboom R, Bos JD, Schmitt J. EASI, (objective) SCORAD and POEM for atopic eczema: responsiveness and minimal clinically important difference. Allergy. 2012 Jan;67(1):99-106. doi: 10.1111/j.1398-9995.2011.02719.x. Epub 2011 Sep 27. PMID 21951293
- [Background] Rausch JR, Maxwell SE, Kelley K. Analytic methods for questions pertaining to a randomized pretest, posttest, follow-up design. J Clin Child Adolesc Psychol. 2003 Sep;32(3):467-86. doi: 10.1207/S15374424JCCP3203_15. PMID 12881035